CLINICAL TRIAL: NCT01747954
Title: Respiratory Mechanics and Hemodynamics in Children With Respiratory Failure: Comparison of Two Techniques of Respiratory Physiotherapy
Brief Title: Effects of Physiotherapy in Hemodynamics and Childrens Respiratory Mechanics
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated
Sponsor: Federal University of Uberlandia (Other)
Responsible Party: Principal Investigator, Letícia de Queiroz Martins, specialist in child health - Clinical Hospital of the Federal University of Uberlândia, Federal University of Uberlandia
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 11112PSC009
Record Dates: First submitted 2012-11-16; First posted 2012-12-12 (Estimated); Last update posted 2012-12-21 (Estimated); Status verified 2012-11

CONDITIONS: Respiratory Insufficiency; Children
Keywords: Respiratory Insufficiency; Physiotherapy Techniques; Respiratory Mechanics
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bag Squeezing (Experimental): * 20% increase in FiO2
  * Inflation pressure of 30 cm H2O + 10l O2/min
  * 0.5 ml saline 0.9%
  * 10 Manual Hyperinflation
  * 10 vibrocompression
  * Aspiration Tracheal
  Interventions: Other: Thoracic vibrocompression
- Thoracic vibrocompression (Active Comparator): * 20% increase in FiO2
  * 0.5 ml saline
  * 10 vibrocompression toracica on the right and left
  * Aspiration Tracheal
  Interventions: Other: Bag Squeezing

INTERVENTIONS:
Other: Bag Squeezing — To perform the BS technique, we used a Protec® manual inflation bag with a flow of 10 L / min and 100% oxygen. A Commercial Medical® manometer was adapted between the orotracheal tube and the inflation bag to monitor the inflation pressure which was recommendedat 30 cmH2O for all children of the BS group. Initially we instilled at most 0.5 ml saline solution(SS) at 0.9% followed by 10 manual hyperinflation maneuvers interspersed with 10 vibrocompression maneuvers and as a last procedure, we performed an aspiration of the orotracheal tube airways and mouth. Between the aspirations the child was re-connected to the ventilator.
  Other Names: BS
  Arms: Thoracic vibrocompression
Other: Thoracic vibrocompression — To perform the TVC technique, we applied 10 vibrocompression maneuvers on the chest of the children during the expiratory phase of the respiratory cycle, on each of the lateral decubitus position, totaling 20 maneuvers, followed by aspiration in the dorsal decubitus position. All measurements in both study groups were performed with the child connected to the ventilator. Before starting the maneuver BS or TVC the child received an increase of 20% fraction of inspired oxygen (FiO2) from what was received previously in MV and after data collection FiO2 returned to baseline values.
  Other Names: TVC
  Arms: Bag Squeezing

SUMMARY:
The hypothesis of this study is that respiratory physiotherapy can promote improvement in respiratory mechanics in children with respiratory failure and the bag squeezing maneuver is more effective in improving respiratory mechanics in childrens and does not alter the hemodynamic proved safe

ELIGIBILITY:
Inclusion Criteria:

* children aged between one and 60 months
* diagnosed with respiratory failure
* undergoing mechanical ventilation

Exclusion Criteria:

* had traumatic brain injury
* severe thrombocytopenia (<20,000 pl/mm³)
* hypovolemia and cyanogenic congenital heart defects
* pneumothorax, hemothorax and/or pleural effusion without previous drainage

Ages: 1 Month to 60 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2010-03; Primary Completion 2011-09 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Effects of Bag Squeezing and vibrocompression chest in hemodynamic, resistance and respiratory system compliance | one hundred twenty minutes
  All variables were assessed prior to the proposed technique (pre-maneuver), immediately after the execution of the technique randomly chosen (post-maneuver), 30, 60 and 120 after the end of the technique randomly chosen. The mean of three readings was used as the representative value for each variable. All children were ventilated with the same mechanical Dixtal® DX3020 Brazil ventilator

SECONDARY OUTCOMES:
comparing all variables between the two groups | one hundred twenty minutes

CONTACTS AND LOCATIONS:
Overall Officials: Letícia Martins, Principal Investigator — Federal University of Uberlandia